

## <u>Patient Consent form – Randomised Controlled Trial</u>

**Study Title:** Developing an arts-based intervention in patients with end-stage kidney disease receiving haemodialysis

Name of Researcher: Claire Carswell

| | | | | Please initial box |
|---|---|---|---|---|
| 1 | I confirm that I have read the information sheet dated 04.07.18, version 0.4 for the above study. I have had the opportunity to consider the information, ask questions, and had my questions answered fully. | | | |
| 2 | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without having my care affected. | | | |
| 3 | I understand that the study is being conducted as part of a PhD project from Queen's University Belfast and that my personal information will be held securely on the university premises and will be handled according to the Data Protection Act 2018 | | | |
| 4 | I understand that data collected as part of this may be looked at by authorized individuals from Queen's University Belfast where it is relevant to my taking part in this research. I give permission for these individuals to have access to this information. | | | |
| 5 | I agree to take part in the above study. | | | |
| Name of participant | | Date | Signature | |
| Researcher | - | | | |
| | | Date | Signature | |
| Anonymous ID code: | | | | |